CLINICAL TRIAL: NCT04889235
Title: Diaphragm Kinetics Following Hepatic Resection, Comparison Between a Sarcopenic and Non-sarcopenic Cohort.
Brief Title: Diaphragm Kinetics Following Hepatic Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Gregory van der Kroft, Principal investigator. Drs., RWTH Aachen University
Other Study IDs: EK 309-18
Record Dates: First submitted 2020-10-21; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Diaphragm Kinetics; Sarcopenia; Muscle Wasting; Liver Resection
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenia: Sarcopenia will be defined as either low estimated muscle mass measured by CT-muscle volumetry or reduced muscle function measured by handgrip strength, or reduced physical condition as defined by the European Working Group on Sarcopenia in Older People (EWGSOP)
  Interventions: Procedure: Major liver resection
- No Sarcopenia: Sarcopenia will be defined as either low estimated muscle mass measured by CT-muscle volumetry or reduced muscle function measured by handgrip strength, or reduced physical condition as defined by the European Working Group on Sarcopenia in Older People (EWGSOP)
  Interventions: Procedure: Major liver resection

INTERVENTIONS:
Procedure: Major liver resection — All patients undergo Major hepatic resection, differences between sarcopenia and no-sarcopenia groups will be observed

SUMMARY:
Sarcopenia is associated with reduced pulmonary function in healthy adults, as well as with increased risk of pneumonia following abdominal surgery. Consequentially, postoperative pneumonia prolongs hospital admission, and increases in-hospital mortality following a range of surgical interventions. Little is known about the function of the diaphragm in the context of sarcopenia and wasting disorders or how its function is influenced by abdominal surgery. Liver surgery induces reactive pleural effusion in most patients, compromising post-operative pulmonary function.

Hypotheses:

* Both major hepatic resection and sarcopenia have a measurable impact on diaphragm function.
* Sarcopenia is associated with reduced preoperative diaphragm function, and that patients with reduced preoperative diaphragm function show a greater decline and reduced recovery of diaphragm function following major hepatic resection.

Goals:

The primary goal of this study is to evaluate whether sarcopenic patients have a reduced diaphragm function prior to major liver resection compared to non-sarcopenic patients, and to evaluate whether sarcopenic patients show a greater reduction in respiratory muscle function following major liver resection when compared to non-sarcopenic patients.

Methods and analysis:

Trans-costal B-mode, M-mode ultrasound and speckle tracking imaging will be used to assess diaphragm function perioperatively in patients undergoing major hepatic resection starting one day prior to surgery and up to thirty days after surgery. In addition, rectus abdominis and quadriceps femoris muscles thickness will be measured using ultrasound to measure sarcopenia, and pulmonary function will be measured using a hand-held bedside spirometer. Muscle mass will be determined preoperatively using CT-muscle volumetry of abdominal muscle and adipose tissue at the third lumbar vertebra level (L3). Muscle function will be assessed using handgrip strength and physical condition will be measured with a short physical performance battery (SPPB). A rectus abdominis muscle biopsy will be taken intraoperatively to measure proteolytic and mitochondrial activity as well as inflammation and redox status. Systemic inflammation and sarcopenia biomarkers will be assessed in serum acquired perioperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18- and 80 years old
* Patients undergoing elective Major hepatic resection for the treatment of malignant disease.
* Patients with all tumor Stages (TNM classification).
* Only patients undergoing Major hepatic resection.

Exclusion Criteria:

* American Anesthesiology Association (ASA)-classification IV or higher
* Liver cirrhosis Child grade B or higher
* End stage renal disease requiring dialysis
* Severe heart disease New York Heart Association class IV
* Pulmonary condition:

  * Chronic obstructive pulmonary disease (COPD)
  * Asthma
  * History of pulmonary surgery
  * History of pulmonary embolism
  * Smoking
  * Pleural effusion occupying more than 1/3 of the pleural space
* Neurological disorders leading to paraparesis of the upper or lower limbs
* Known muscular dystrophic disorders

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will entail a prospective observational single center study, analyzing 44 consecutive patients undergoing major liver resection, 22 patients will be sarcopenic, 22 will be non-sarcopenic
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Diaphragm kinetics | Day 1
  Comparing diaphragm kinetics between sarcopenic and non-sarcopenic patients prior to elective major hepatic resection using ST ultrasound.
  Diaphragm muscle kinetics will be evaluated using the following outcome value.
  -Deformation%
  Mean values and standard deviations of individual values describing diaphragm kinetics of sarcopenic and non-sarcopenic groups will be compared. Preoperative values will be used as baseline values for the evaluation of longitudonal changes (secondary outcome measure)
Diaphragm kinetics | Day 1
  Comparing diaphragm kinetics between sarcopenic and non-sarcopenic patients prior to elective major hepatic resection using ST ultrasound.
  Diaphragm muscle kinetics will be evaluated using the following value.
  -Deformation velocity (in cm/second)
  Mean values and standard deviations of individual values describing diaphragm kinetics of sarcopenic and non-sarcopenic groups will be compared. Preoperative values will be used as baseline values for the evaluation of longitudonal changes (secondary outcome measure)
Diaphragm kinetics | Day 1
  Comparing diaphragm kinetics between sarcopenic and non-sarcopenic patients prior to elective major hepatic resection using ST ultrasound.
  Diaphragm muscle kinetics will be evaluated using the following value.
  -Fractional thickening (thickening coefficient)
  Mean values and standard deviations of individual values describing diaphragm kinetics of sarcopenic and non-sarcopenic groups will be compared. Preoperative values will be used as baseline values for the evaluation of longitudonal changes (secondary outcome measure)
Diaphragm kinetics | Day 1
  Comparing diaphragm and abdominal muscle kinetics between sarcopenic and non-sarcopenic patients prior to elective major hepatic resection using ST ultrasound.
  Diaphragm muscle kinetics will be evaluated using the following value.
  -Range of DIA (in cm)
  Mean values and standard deviations of individual values describing diaphragm kinetics of sarcopenic and non-sarcopenic groups will be compared. Preoperative values will be used as baseline values for the evaluation of longitudonal changes (secondary outcome measure)
Abdominal muscle kinetics | Day 1
  Primary outcome:
  Comparing abdominal muscle kinetics between sarcopenic and non-sarcopenic patients prior to elective major hepatic resection using ST ultrasound.
  Abdominal muscle kinetics will be evaluated using the following value.
  -Thickness (in cm)
  Mean values and standard deviations of individual values describing abdominal muscle kinetics of sarcopenic and non-sarcopenic groups will be compared. Preoperative values will be used as baseline values for the evaluation of longitudonal changes (secondary outcome measure)
Abdominal muscle kinetics | Day 1
  Primary outcome:
  Comparing abdominal muscle kinetics between sarcopenic and non-sarcopenic patients prior to elective major hepatic resection using ST ultrasound.
  Abdominal muscle kinetics will be evaluated using the following value.
  -Deformation%
  Mean values and standard deviations of individual values describing abdominal muscle kinetics of sarcopenic and non-sarcopenic groups will be compared. Preoperative values will be used as baseline values for the evaluation of longitudonal changes (secondary outcome measure)
Abdominal muscle kinetics | Day 1
  Primary outcome:
  Comparing abdominal muscle kinetics between sarcopenic and non-sarcopenic patients prior to elective major hepatic resection using ST ultrasound.
  Abdominal muscle kinetics will be evaluated using the following value.
  -Deformation velocity (in cm/second)
  Mean values and standard deviations of individual values describing abdominal muscle kinetics of sarcopenic and non-sarcopenic groups will be compared. Preoperative values will be used as baseline values for the evaluation of longitudonal changes (secondary outcome measure)

SECONDARY OUTCOMES:
Diaphragm kinetics | 30 days
  Evaluating longitudinal changes in diaphragm kinetics in the postoperative phase across sarcopenic and non-sarcopenic groups following elective major hepatic resection using ST ultrasound.
  Diaphragm muscle kinetics will be evaluated using the following value.
  -Deformation%
  Differences in mean values and standard deviations of individual values describing diaphragm muscle kinetics will be compared between sarcopenic and non-sarcopenic groups. Changes in diaphragm kinetics will be defined as changes from baseline values (primary outcome).
Diaphragm kinetics | 30 days
  Evaluating longitudinal changes in diaphragm kinetics in the postoperative phase across sarcopenic and non-sarcopenic groups following elective major hepatic resection using ST ultrasound.
  Diaphragm muscle kinetics will be evaluated using the following value.
  -Deformation velocity (in cm/second)
  Differences in mean values and standard deviations of individual values describing diaphragm muscle kinetics will be compared between sarcopenic and non-sarcopenic groups. Changes in diaphragm kinetics will be defined as changes from baseline values (primary outcome).
Diaphragm kinetics | 30 days
  Evaluating longitudinal changes in diaphragm kinetics in the postoperative phase across sarcopenic and non-sarcopenic groups following elective major hepatic resection using ST ultrasound.
  Diaphragm muscle kinetics will be evaluated using the following value.
  -Fractional thickening (thickening coefficient)
  Differences in mean values and standard deviations of individual values describing diaphragm muscle kinetics will be compared between sarcopenic and non-sarcopenic groups. Changes in diaphragm kinetics will be defined as changes from baseline values (primary outcome).
Diaphragm kinetics | 30 days
  Evaluating longitudinal changes in diaphragm kinetics in the postoperative phase across sarcopenic and non-sarcopenic groups following elective major hepatic resection using ST ultrasound.
  Diaphragm muscle kinetics will be evaluated using the following value.
  -Range of DIA (in cm)
  Differences in mean values and standard deviations of individual values describing diaphragm muscle kinetics will be compared between sarcopenic and non-sarcopenic groups. Changes in diaphragm kinetics will be defined as changes from baseline values (primary outcome).
Abdominal muscle kinetics | 30 days
  Evaluating longitudinal changes in abdominal muscle kinetics in the postoperative phase across sarcopenic and non-sarcopenic groups following elective major hepatic resection using ST ultrasound.
  Abdominal muscle kinetics will be evaluated using the following value.
  -Thickness (in cm)
  Differences in mean values and standard deviations of individual values describing abdominal muscle kinetics will be compared between sarcopenic and non-sarcopenic groups. Changes in diaphragm kinetics will be defined as changes from baseline values (primary outcome).
Abdominal muscle kinetics | 30 days
  Evaluating longitudinal changes in abdominal muscle kinetics in the postoperative phase across sarcopenic and non-sarcopenic groups following elective major hepatic resection using ST ultrasound.
  Abdominal muscle kinetics will be evaluated using the following value.
  -Deformation%
  Differences in mean values and standard deviations of individual values describing abdominal muscle kinetics will be compared between sarcopenic and non-sarcopenic groups. Changes in diaphragm kinetics will be defined as changes from baseline values (primary outcome).
Abdominal muscle kinetics | 30 days
  Evaluating longitudinal changes in abdominal muscle kinetics in the postoperative phase across sarcopenic and non-sarcopenic groups following elective major hepatic resection using ST ultrasound.
  Abdominal muscle kinetics will be evaluated using the following value.
  -Deformation velocity (in cm/second)
  Differences in mean values and standard deviations of individual values describing abdominal muscle kinetics will be compared between sarcopenic and non-sarcopenic groups. Changes in diaphragm kinetics will be defined as changes from baseline values (primary outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Uniklinik Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No